CLINICAL TRIAL: NCT00253279
Title: A Quantitative Study of the Metabolic Alterations in Protein Synthesis Rate That Occur in Burn Patients Over the Time Course of Their Injury Using Positron Emission Tomography.
Brief Title: Alterations in Protein Synthesis Rates of Burn Patients Measured Over Time Using PET Scans
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Ronald G. Tompkins, MD, ScD, Chief, Burn Service, Massachusetts General Hospital
Organization: National Institute of General Medical Sciences (NIGMS) (NIH)
Other Study IDs: 2005-P-001510; G P50 GM021700-28
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2009-08-13 (Estimated); Status verified 2009-08

CONDITIONS: Burn
Keywords: Protein Synthesis Rate; Burn Injury; PET Scan
MeSH Terms: conditions — Burns | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: 16 healthy subjects will be studied. Each patient will undergo one PET Scan to measure muscle protein synthesis rate.
  Interventions: Procedure: PET Scans
- 2: 48 burn patients will be studied. Each patient will have a maximum of 3 PET Scans, which will be done at different times during the first 24 months after injury. A maximum of 2 of these scans will be done while they are inpatient; one after discharge.
  Interventions: Procedure: PET Scans

INTERVENTIONS:
Procedure: PET Scans — Healthy volunteers will undergo one PET Scan; bur patients will undergo a maximum of 3 PET scans over 2 years after injury; a maximum of 2 will be done while inpatient; one after d/c.
  Other Names: PET Scan; Muscle Protein Metabolism

SUMMARY:
Our specific aim is to gain an understanding of protein synthesis rates in burn patients at various times during their injury and recovery by using PET scans. This will be compared with healthy volunteer controls. We hope this will help optimize nutrition and care regimens for future burn patients.

DETAILED DESCRIPTION:
The purpose of this study is to understand how muscles are built up and broken down (metabolism) in both burn patients and healthy people.The studies will help us understand how muscle metabolism is different for burn patients and healthy subjects. We hope to find ways to help the body of a burn victim heal without losing too much muscle.

Protein is an important part of our daily diet. Normally, the body breaks down the protein we eat into smaller pieces called amino acids. It uses the amino acids to make its own proteins. It uses these proteins to heal wounds, fight infections, and provide energy.

After a burn injury, the body speeds up the pace of its life activities. It needs more energy just to stay alive and recover from the burn. The body often gets the extra energy it needs by breaking the protein in muscles down into amino acids. The amino acids are then made into new proteins. If too much muscle is broken down, it is harder for the body to function. This can make recovery slower or possibly lead to death.

For Healthy Volunteers, this study will require no more than 6 hours of time in total. This time will be spread out over two visits, a Screening Visit and a Scan Visit.

For Burn Patients, this study will require no more than 14 hours total. This time will be spread out over four visits-a screening visit and a maximum of 3 scan visits. A total of three PET scans will be done over a 2 year period.

ELIGIBILITY:
Inclusion Criteria:

FOR HEALTHY VOLUNTEERS

Healthy males and females 18-70 years of age.

Laboratory results within MGH-accepted normal range.

Within 20% of the ideal weight for their height.

Supine and standing blood pressure within the range of 110/60 to 150/90 mm Hg

Heart rate within the range of 46-90 beats/minute after 5 minutes of rest.

Subjects <40 years old with HCT >=24, age 40-60 with HCT >=27, age 60-70 with HCT >=30.

FOR BURN SUBJECTS:

Inclusion Criteria:

Burn Injury of >=5 % TBSA from any cause.

18 -70 years of age

Stable hemodynamic and cardiopulmonary states as judged by the attending surgeons in the burn unit.

Patient who is capable of giving full informed consent.

Exclusion Criteria:

FOR HEALTHY SUBJECTS Clinical evidence of physical or mental disease.

Clinically significant abnormality of the laboratory tests.

Known drug or alcohol dependence.

History of drug allergy

Taking standard prescription drugs within two weeks or investigational drugs within four weeks prior to the PET scan

Diabetes mellitus and other metabolic endocrine disorders Pregnant or lactating

FOR BURN SUBJECTS:

Pregnant or lactating females

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects and burn patients
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald T Tompkins, MD, ScD, Principal Investigator — Massachusetts General Hospital, Shriners Burn Hospital- Boston
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Fischman AJ, Hsu H, Carter EA, Yu YM, Tompkins RG, Guerrero JL, Young VR, Alpert NM. Regional measurement of canine skeletal muscle blood flow by positron emission tomography with H2(15)O. J Appl Physiol (1985). 2002 Apr;92(4):1709-16. doi: 10.1152/japplphysiol.00445.2001. PMID 11896041
- [Background] Fischman AJ, Yu YM, Livni E, Babich JW, Young VR, Alpert NM, Tompkins RG. Muscle protein synthesis by positron-emission tomography with L-[methyl-11C]methionine in adult humans. Proc Natl Acad Sci U S A. 1998 Oct 27;95(22):12793-8. doi: 10.1073/pnas.95.22.12793. PMID 9788993
- [Background] Hsu H, Yu YM, Babich JW, Burke JF, Livni E, Tompkins RG, Young VR, Alpert NM, Fischman AJ. Measurement of muscle protein synthesis by positron emission tomography with L-[methyl-11C]methionine. Proc Natl Acad Sci U S A. 1996 Mar 5;93(5):1841-6. doi: 10.1073/pnas.93.5.1841. PMID 8700846
- [Background] Carter EA, Yu YM, Alpert NM, Bonab AA, Tompkins RG, Fischman AJ. Measurement of muscle protein synthesis by positron emission tomography with L-[methyl-11C]methionine: effects of transamination and transmethylation. J Trauma. 1999 Aug;47(2):341-5. doi: 10.1097/00005373-199908000-00021. PMID 10452471